CLINICAL TRIAL: NCT02831322
Title: A Study of Structure and Function of Radial Artery After Transradial Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21735
Record Dates: First submitted 2016-07-04; First posted 2016-07-13 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Intervention; Transradial
Keywords: Transradial; ﬂow-mediated vasodilation
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- radial artery occlusion (Experimental): Radial artery occlusion was the absence of a flow signal by Doppler ultrasound examination.
  Interventions: Procedure: Percutaneous coronary intervention
- radial artery normal (Other): Radial artery normal was blood flow signal by Doppler ultrasound
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention was a nonsurgical technique for treating obstructive coronary artery disease

SUMMARY:
Several approaches have been proposed to reduce the risk of RAO, including anticoagulation, immediate postprocedural sheath removal, and a small sheath/radial artery ratio. Doppler ultrasound examination showed that interrupted blood flow in RA tend to occur in the proximal end rather than distal part of the artery,which was ignored by a majority of interventional cardiologists. Different insights into occlusion location may lead to different options of sheath materials, models, catheters and puncture access. Thus, the investigators designed this present study to explore the reason of radial artery endothelial dysfuction and damage and occlusion location by ﬂow-mediated dilation (FMD) to determine the suitable method to reduce occlusion risk during TRI.

ELIGIBILITY:
Inclusion Criteria:

* admitted for transradial catheterization.

Exclusion Criteria:

* femoral access, arterial circulatory disease, pathological Allen tests, decompensated heart failure, chronic renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
radial artery occlusion | 6 month
  radial artery occlusion was the absence of a flow signal by Doppler ultrasound examination

CONTACTS AND LOCATIONS:
Locations (1):
- Qingsheng wang, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes